CLINICAL TRIAL: NCT01469273
Title: Prophylaxis of Gastrointestinal Infections in Newborn and Infants With a Suspension Containing the Probiotic Escherichia Coli Strain Nissle
Brief Title: Prophylaxis of Gastrointestinal Infections With EcN
Acronym: PIURA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital San Bartolome (Other)
Collaborators: Instituto de Investigacion de las Alteraciones del Crecimiento, Desarrollo y Enfermedades Metabolicas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MU 0932 BL
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Infantile Diarrhea
Keywords: Diarrhea; EcN; E. coli strain Nissle 1917; Gastrointestinal infection; Infant; Newborn; Probiotic drug; Prevention; Prophylaxis
MeSH Terms: conditions — Diarrhea, Infantile; Diarrhea | interventions — 17-hydroxyestrane-3-carbonitrile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): Only observation; observation period: 1 year.
- Early Treatment group (E) (Experimental): 1 x 1 ml of EcN suspension/day on 10 consecutive days, application in the morning before feeding/nursing, first application 48h after birth, latest. Observation period: 1 year.
  Interventions: Drug: Mutaflor® Suspension
- Late Treatment Group (L) (Experimental): 1 x 1 ml of EcN suspension/day on 10 consecutive days, application in the morning after feeding/nursing, starting on the first day of the 7th month of life. Observation period: 1 year.
  Interventions: Drug: Mutaflor® Suspension

INTERVENTIONS:
Drug: Mutaflor® Suspension — Application of Mutaflor-Suspension on 10 consecutive days.
  Other Names: EcN; Mutaflor; Newborn; Nissle; Prophylaxis
  Arms: Early Treatment group (E); Late Treatment Group (L)

SUMMARY:
This interventional trial shall investigate the efficacy and tolerance of a suspension with non-pathogenic probiotic E. coli strain Nissle (EcN) on prophylaxis against gastrointestinal infections in newborn and infants. ECN-SUSPENSION is a probiotic containing viable E. coli bacteria of the non-pathogenic Nissle 1917 strain at a concentration of 10exp8 cells per ml.

DETAILED DESCRIPTION:
Newborns (treatment-group E) and infants at the age of 6 months (treatment-group L) shall be treated with 1 x 1 ml ECN-SUSPENSION for 10 days and observed until the age of 12 months.Treatment-group E (newborn) will receive EcN-Suspension on the first 10 days of life and will be observed for the next 12 months. Treatment-group L (infants at the age of 6 months) will receive EcN-Suspension on the first 10 days of their seventh month of life and will be observed for the next 6 months.The corresponding control group will remain untreated and will be observed only for 12 months. According to the hospitals daily routine the inclusion and exclusion criteria will be checked. All newborns meeting the inclusion criteria will be included into the trial. Patients' anamnestic data and general health status are recorded at the initial control.Controls are performed according to the time schedule normally used in the hospital functioning as a trial site. According to this, during each monthly control data on the efficacy and safety are recorded. The final control for assessing the tolerance and efficacy of the trial medication is conducted along with a physical examination after an observation period of 12 months.In this study, diarrhea is defined as increase of stool frequency to >3 watery or loose stools in 24 hours on at least two or more consecutive days.The prophylaxis against gastrointestinal infections with EcN-Suspension is expected to result in a decrease of the number episodes of diarrhea in comparison to the untreated control. The primary efficacy criterion is the number of episodes of diarrhea caused by gastrointestinal infection within the first 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed by the patient's parents or legal guardians.
* Term born infants.

  * Age < 2 days
  * Gestational age from 38-42 weeks of gestation
  * Birth weight from 2500-3750 gr.
  * Normal delivery (eutocia)

Exclusion criteria:

* Simultaneous participation in another clinical study
* Consumption of food supplements or medicines containing live micro-organisms or their metabolic products or components during the study
* Other reasons which in the opinion of the investigator provide a reason against the inclusion of the patient in the study.
* Autoimmune disease·Severe sepsis or severe systemic injury
* Immunosuppressive treatment
* Severe co-morbidities diseases of the:

  * Heart
  * Liver
  * Kidney
* Genetic disease
* Other serious associated diseases, which in the opinion of the investigator, cast a doubt on the implementation of the test according to the study protocol.

Ages: 3 Hours to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 198 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Number of diarrhea episodes | 12 months / first year of life
  To show superiority of a prophylaxis with a probiotic suspension containing E. coli strain Nissle against gastrointestinal infections associated with diarrhea, compared to an untreated control group

SECONDARY OUTCOMES:
Number of days with diarrhea | 12 months / first year of life
  To show prophylaxis with a probiotic suspension containing E. coli strain Nissle against gastrointestinal infections associated with diarrhea within the first 12 months of life compared to an untreated control group.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Bindels, MD, Principal Investigator — Hospital San Bartolome
Locations (3):
- Peru (3):
  - Centro de Salud Los Algarrobos, Piura, Piura
  - Centro de Salud Materno Inftantil de Castilla (CESAMICA), Piura, Piura
  - Materno Infantil Santa Rosa, Piura, Piura